CLINICAL TRIAL: NCT02240225
Title: Validation of Chinese Severe Respiratory Insufficiency （SRI）Questionnaire for COPD Patients With Chronic Hypercapnic Respiratory Failure
Brief Title: Validation of Chinese SRI Questionnaire
Acronym: VCSRI
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Guangzhou Institute of Respiratory Disease (Other)
Collaborators: Southern Medical University, China (Other); Second Affiliated Hospital, Sun Yat-Sen University (Other); Third Affiliated Hospital, Sun Yat-Sen University (Other); Shaoguan People's Hospital (Unknown); Dongguan People's Hospital (Other Government); The center hospital of Wuhan (Unknown)
Responsible Party: Principal Investigator, LuQian Zhou, Assistant professor of Guangzhou Institute of Respiratory Disease, Guangzhou Institute of Respiratory Disease
Other Study IDs: GZIRD-20140910
Record Dates: First submitted 2014-09-11; First posted 2014-09-15 (Estimated); Last update posted 2014-09-15 (Estimated); Status verified 2014-09

CONDITIONS: Chronic Obstructive Pulmonary Disease; Hypercapnic Respiratory Failure
Keywords: COPD;SRI;Reliability;validity;
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Respiratory Insufficiency

STUDY DESIGN:
Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Weeks
Oversight: Data Monitoring Committee: No

SUMMARY:
Assessment of health-related quality of life in COPD patients with severe chronic respiratory failure requires appropriate and highly specific measurement tools. We attempt to validate the Chinese version of the Severe Respiratory Insufficiency Questionnaire (SRI)

ELIGIBILITY:
Inclusion Criteria:

1. Adult COPD Patients with chronic hypercapnic respiratory failure established on home noninvasive ventilation for at least 1 month
2. Patients are in a clinically stable state,without any changes of medication during the previous 4 weeks.

Exclusion Criteria:

1. patient's refusal to participate
2. Patients with evidence of acute respiratory failure i.e.patients with worsening of symptoms during the previous 2 weeks, a pH ,7.35, or with signs of respiratory infection

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult COPD patients with chronic hypercapnic respiratory failure receiving home noninvasive ventilation
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2014-01; Primary Completion 2014-10 (Estimated); Study Completion 2014-10 (Estimated)

PRIMARY OUTCOMES:
Reliability of Severe Respiratory Insufficiency Questionnaire | 2 weeks

SECONDARY OUTCOMES:
Construct validity of Severe Respiratory Insufficiency Questionnaire | 2 weeks
Criterion validity of Severe Respiratory Insufficiency Questionnaire | 2 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Guangzhou Institute of Respiratory Disease, Guangzhou, Guangdong, China